CLINICAL TRIAL: NCT01951872
Title: Treatment for Caffeine Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00051415; R01DA003890 (NIH)
Record Dates: First submitted 2013-09-20; First posted 2013-09-27 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Caffeine Use Disorder (DSM-5 Condition for Further Study)
Keywords: caffeine dependence; caffeine withdrawal; caffeine use disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (Experimental): Immediate manual-based treatment for caffeine dependence: administered within approximately one week following intake.
  Interventions: Behavioral: Manual-based treatment for caffeine dependence
- Delayed treatment (Experimental): Delayed manual-based treatment for caffeine dependence: administered within approximately six weeks following intake.
  Interventions: Behavioral: Manual-based treatment for caffeine dependence

INTERVENTIONS:
Behavioral: Manual-based treatment for caffeine dependence — Participants will meet with a counselor to discuss plans for caffeine reduction or cessation, and they will receive a manual-based treatment to help guide them through caffeine reduction or cessation.

SUMMARY:
Recent research has shown that some individuals become addicted to or dependent on caffeine and are unable to quit or reduce caffeine consumption despite a persistent desire to do so. The aims of the current study are to characterize caffeine use among individuals with physical or psychological dependence on caffeine and evaluate a manual-based intervention to promote caffeine reduction and cessation.

DETAILED DESCRIPTION:
A large percentage of caffeine users in the general population (56%) report a persistent desire or unsuccessful efforts to stop or reduce caffeine consumption. The aim of Study 1 is to recruit and identify individuals who are interested in receiving treatment to reduce or quit caffeine consumption. Individuals will be recruited from Baltimore, MD and surrounding communities via flyers and newspaper and radio advertisements. Those who are eligible will be invited to come to the Behavioral Pharmacology Research Unit located on the Johns Hopkins Bayview Medical Center campus in Baltimore, MD. After consent is obtained at intake (consent form A), a series of questionnaires will be completed (e.g., demographics, caffeine history, medical and psychiatric history, mood), followed by a structured clinical interview that will assess caffeine use and dependence. Individuals who meet eligibility criteria will be offered the opportunity to receive assistance to reduce or quit caffeine. Those who consent (consent form B) to enroll in the second phase of the project will be randomly assigned to one of two conditions: 1) immediate treatment or 2) delayed treatment. The conditions will be identical with the exception of a 6 week delay for the delayed treatment group. Participants will receive a caffeine reduction and cessation treatment manual during a brief treatment session at week 1. Treatment progress will be assessed during a study session approximately 7 weeks post-treatment, during a telephone interview approximately 8 weeks post-treatment, and during a follow-up telephone call approximately 27 weeks after the treatment session. Progress will be assessed via questionnaires, food diaries, and salivary caffeine measures.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy
* Self-reported problem with caffeine use
* Moderate to heavy caffeine use

Exclusion Criteria:

* Pregnancy
* Current dependence on alcohol or illicit drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in self-reported caffeine use | Measure will be assessed at weeks 1, 7, 8, and 27.

SECONDARY OUTCOMES:
Change in biological measure of caffeine use | Measure will be assessed at weeks 1 and 7.
  Salivary caffeine

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Griffiths, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States